CLINICAL TRIAL: NCT02241395
Title: Autologous Bone Marrow Mononuclear Cell Therapy in Cerebral Palsy
Brief Title: Cell Therapy as Treatment for Cerebral Palsy
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Neurogen Brain and Spine Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NGBSI-09
Record Dates: First submitted 2014-09-12; First posted 2014-09-16 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; autologous bone marrow mononuclear cells; stem cell
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stem Cell (Experimental): Intrathecal autologous bone marrow mononuclear cell transplantation
  Interventions: Biological: Intrathecal autologous bone marrow mononuclear cell transplantation

INTERVENTIONS:
Biological: Intrathecal autologous bone marrow mononuclear cell transplantation

SUMMARY:
The purpose of this study was to study the effect of autologous bone marrow mononuclear cells on common symptoms of cerebral palsy patients.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed cases of any type of Cerebral Palsy
* age above 6 months.

Exclusion Criteria:

* presence of acute infections such as Human immunodeficiency virus/Hepatitis B Virus/ Hepatitis C Virus
* malignancies
* bleeding tendencies
* pneumonia
* renal failure
* severe liver dysfunction
* severe anemia [Hemoglobin < 8]
* any bone marrow disorder
* space occupying lesion in brain
* other acute medical conditions such as respiratory infection and pyrexia.

Ages: 6 Months to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2013-08; Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
change in clinical symptoms over a period of 2 years | 2 years
  Clinical symptoms such as oromotor skills, sitting and standing balance, speech, ambulation, muscle tone, cognition, hand and leg movement, walking, etc

SECONDARY OUTCOMES:
Change in GMFM score | 1 year
Change in Gross Motor Function Measure | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Neurogen brain and spine institute, Navi Mumbai, Maharashtra, India